CLINICAL TRIAL: NCT06632392
Title: The Effect of Simulation-Based Preoperative Nursing Care Education on Student Anxiety and Competence in Care
Brief Title: The Effect of Simulation-Based Preoperative Nursing Care Education on Student
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Niran Coban, Asst.Prof.Dr., Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BYZ
Record Dates: First submitted 2024-10-06; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Preoperative Care; Nursing Education; Simulation; Clinical Practice

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theory and simulation training (Experimental): I. Interview: Before theoretical and simulation training II. Interview: After theoretical and simulation training III. Interview: Four weeks later
  Interventions: Other: Simulation training; Other: Theory training
- Standart Theory training (Other): I. Interview: Before theoretical and simulation training II. Interview: After theoretical training III. Interview: Four weeks later
  Interventions: Other: Theory training

INTERVENTIONS:
Other: Simulation training — Theory and simulation training
  Arms: Theory and simulation training
Other: Theory training — Theory training

SUMMARY:
Today, different technologies are used in the stages of the education and training process. Simulation education approaches constitute an important group in health education and training. Simulation in nursing education; provides experience-based learning opportunities and enables students to develop their clinical decision-making skills. The aim of this study is to determine the competence status and influencing factors of students who continue their nursing education at the faculty of health sciences of a foundation university regarding preoperative nursing care. This randomized controlled study will be conducted with students who continue their nursing education at the faculty of health sciences at a foundation university on the Anatolian side of Istanbul in the 2023-2024 academic year. The research data were obtained with an introductory questionnaire, Perceived Competence Scale for Preoperative Nursing Care, Kolb Learning Styles Inventory III, STAI State and Trait Anxiety Scale. Before the data collection process, Ethics Committee approval and institutional permission were obtained, the purpose of the study was explained to the students and an informed consent form was filled out. Students who agreed to participate in the study filled out the relevant survey questionnaires and scale questions. The aim of this study is to determine the effect of simulation-based education to be given to nursing students on their perceived competence status and anxiety levels regarding preoperative nursing care. This randomized controlled study will shed light on future studies.

ELIGIBILITY:
Inclusion Criteria:

* -2023-2024 Students actively continuing their undergraduate nursing program at the Faculty of Health Sciences
* Students who volunteered to participate in the research were included in the research

Exclusion Criteria:

* Students who have graduated
* Those who did not volunteer were not included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The effects of simulation and theory training on preoperative nursing care competencies of students. | 4 week
  Perceived Competence Scale for Preoperative Nursing Care: It was created in line with the nursing competencies published by the International Council of Nurses and the perioperative period nursing practice competencies presented by the European Association of Operating Theatre Nurses and a comprehensive literature review. This scale was designed to support nurses to receive a competency-based training in order to fulfil their responsibilities in preoperative care in the most effective way and to measure their competencies during the training process. The scale consists of five sub-dimensions and includes 22 questions in total.
The effects of simulation and theory training on students' anxiety levels | 4 week
  State Anxiety Inventory: In our study, the "State Anxiety Inventory" will be used before and after the procedure to evaluate the anxiety levels of the patients in a certain situation.The "State Anxiety Inventory (STAI-I)" is a tool that measures how the individual feels at a particular moment and situation, that is, the level of anxiety in that condition. Post-Surgery - After Transfer to the Clinic: Before the Su Jok application, the patient's anxiety status will be determined by the State-Trait Anxiety Inventory (STAI-I),For 30 minutes, the point where the seed is fixed will be massaged with the Su Jok technique,15 minutes after the Su Jok application, the patient's pain status will be determined by the State-Trait Anxiety Inventory (STAI-I).These stages will be applied again on the 1st and 2nd days after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Niran çoban, Asist. Prof., Study Director — Okan University
Locations (1):
- Istanbul- City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Terzioglu F, Yucel C, Koc G, Simsek S, Yasar BN, Sahan FU, Akin R, Ocal SE, Akdag C, Elcin M, Mert M, Yildirim S. A new strategy in nursing education: From hybrid simulation to clinical practice. Nurse Educ Today. 2016 Apr;39:104-8. doi: 10.1016/j.nedt.2016.01.009. Epub 2016 Jan 28. PMID 27006040
- [Background] Simsek P, Ozmen GC, Kemer AS, Aydin RK, Bulut E, Cilingir D. Development and psychometric testing of Perceived Preoperative Nursing Care Competence Scale for Nursing Students (PPreCC-NS). Nurse Educ Today. 2023 Jan;120:105632. doi: 10.1016/j.nedt.2022.105632. Epub 2022 Nov 11. PMID 36410082
- [Background] Durmaz Edeer A, Vural F, Turhan Damar H, Yasak K, Damar M. The Effect of Web-Based Preoperative and Postoperative Patient Care Education on Nursing Students: A Randomized Controlled Study. Comput Inform Nurs. 2019 Oct;37(10):541-547. doi: 10.1097/CIN.0000000000000552. PMID 31373901